CLINICAL TRIAL: NCT00243087
Title: An Open Phase I Single Dose Escalation Study of BI 2536 Administered Intravenously in Patients With Refractory or Relapsed Non-Hodgkin's Lymphoma
Brief Title: Investigation of Safety, Tolerability and Maximum Tolerated Dose (MTD) of BI 2536 in Patients With Recurrent Advanced Aggressive Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000446176; BOEH-BI-1216.3; UNMC-16005
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Lymphoma
Keywords: stage IV adult diffuse large cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; stage IV grade 3 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; anaplastic large cell lymphoma; recurrent adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult T-cell leukemia/lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Large-Cell, Anaplastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — BI 2536

INTERVENTIONS:
Drug: BI 2536

SUMMARY:
RATIONALE: BI 2536 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of BI 2536 in treating patients with refractory or relapsed advanced non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of BI 2536 in patients with refractory or relapsed advanced aggressive non-Hodgkin's lymphoma.
* Determine the safety and tolerability of this drug in these patients.

Secondary

* Determine the pharmacokinetic profile of this drug in these patients.
* Determine, preliminarily, the antitumor activity of this drug in these patients.

OUTLINE: This is a dose-escalation, open-label, uncontrolled, multicenter study.

Patients receive BI 2536 IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BI 2536 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity during the first treatment course. Up to 24 patients are treated at the MTD.

After completion of study treatment, patients are followed periodically until disease progression or initiation of another cancer treatment.

PROJECTED ACCRUAL: A maximum of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced aggressive non-Hodgkin's lymphoma (NHL), including any of the following subtypes:

  * B-cell NHL, including any of the following subtypes:

    * Diffuse large B-cell lymphoma
    * Primary mediastinal (thymic) B-cell lymphoma
    * Intravascular large B-cell lymphoma
    * Immunoblastic B-cell lymphoma
    * Mantle cell lymphoma
    * Burkitt's lymphoma
    * Follicular grade 3b lymphoma
  * T-cell NHL, including any of the following subtypes:

    * Anaplastic large cell lymphoma
    * Peripheral T-cell lymphoma, not otherwise specified
* De novo or transformed disease
* Refractory (i.e., disease not amenable to standard therapy) or relapsed disease, as evidenced by 1 of the following:

  * Refractory to OR relapsed after ≥ 1 prior combination chemotherapy regimen
  * Refractory to OR relapsed after prior CD20-based immunotherapy (for patients eligible to receive such therapy)
  * Refractory after prior high-dose chemotherapy and autologous stem cell transplantation AND ≥ 100 days post transplantation
* At least 1 bidimensionally measurable lesion ≥ 1.5 cm by CT scan, MRI, x-ray, or clinical examination
* No active CNS lymphoma

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 9 g/dL
* No known coagulopathy

Hepatic

* ALT and/or AST ≤ 2.5 times upper limit of normal (ULN) (< 5 times ULN if due to hepatic lymphoma)
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 2.0 mg/dL

Immunologic

* No known HIV infection
* No serious active infection that requires IV antibiotics or antifungal or antiviral agents

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception during and for 1 year after completion of study treatment
* No known or suspected alcohol or drug abuse
* No sensory or motor neuropathy ≥ grade 3
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No other life-threatening illness or organ dysfunction that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* See Radiotherapy
* More than 3 weeks since prior and no concurrent immunotherapy
* No prior allogeneic bone marrow transplantation

Chemotherapy

* See Disease Characteristics
* More than 3 weeks since prior and no concurrent chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy

* No concurrent hormonal therapy

Radiotherapy

* No prior radiotherapy to the only site of measurable disease unless there is documented disease progression after completion of radiotherapy
* More than 8 weeks since prior and no concurrent systemic radioimmunotherapy
* More than 3 weeks since prior and no concurrent radiotherapy

  * Concurrent palliative radiotherapy to sites other than the only measurable target lesion allowed for symptom control provided the reason for radiotherapy does not reflect progressive disease

Other

* No concurrent warfarin for therapeutic anticoagulation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-07; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose as measured by CTCAE v3.0 at days 1-22 of each course | up to 22 days of each course
Dose-limiting toxicity as measured by CTCAE v3.0 at days 1-22 of each course | up to 22 days of each course

SECONDARY OUTCOMES:
Objective tumor response by CT scan or MRI as measured by RECIST criteria on day 22 of each even numbered course | day 22 of every second course
Pharmacokinetics as measured in blood samples at days 1, 2, 3, and 8 during first course and on day 1 of each subsequent course | day 22 of each course

CONTACTS AND LOCATIONS:
Overall Officials: Julie M. Vose, MD, Study Chair — University of Nebraska
Locations (4):
- United States (4):
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing